CLINICAL TRIAL: NCT01686009
Title: Intra-nasal Ketamine for Analgesia in the Emergency Department
Acronym: INKA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Lions Gate Hospital (Other)
Collaborators: North Shore Health Research Foundation (Unknown)
Responsible Party: Principal Investigator, Gary Andolfatto, Assistant Professor, University of British Columbia Department of Emergency Medicine; Attending Physician and Emergency Department Research Director, Lions Gate Hospital, Lions Gate Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UBC Dept of EM
Record Dates: First submitted 2012-09-12; First posted 2012-09-17 (Estimated); Last update posted 2013-02-05 (Estimated); Status verified 2013-02

CONDITIONS: Pain
Keywords: pain; analgesia; ketamine; intranasal; emergency
MeSH Terms: conditions — Pain; Agnosia; Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intra-nasal ketamine (Experimental): 0.5 mg/kg ketamine intra-nasally; then 0.25 mg/kg repeat dose after 10 minutes if necessary
  Interventions: Drug: Intra-nasal ketamine

INTERVENTIONS:
Drug: Intra-nasal ketamine

SUMMARY:
The provision of analgesia to patients in pain is a fundamental necessity of emergency department practice and is usually accomplished using IV opioids. However, significant barriers exist to the provision of timely analgesia by the IV route.

The use of the IN route for medication delivery provides an efficient and relatively painless mode of analgesia delivery. As well, ketamine is well-known to be an effective analgesic and to preserve cardiorespiratory function thus removing the necessity of physiologic monitoring that is obligatory when using opioids. The use of ketamine by the IN route provides a rapid, easy-administered and well-tolerated method for providing analgesia in the ED setting.

ELIGIBILITY:
Inclusion Criteria:

* age 6 years or greater
* moderate or severe pain (VAS >=50mm)

Exclusion Criteria:

* history of allergy or intolerance to ketamine
* structural or functional nasal occlusion
* inability to understand the VAS
* Glasgow Coma Scale < 15
* Systolic BP > 180
* History of schizophrenia
* Clinical necessity for immediate IV access as judged by the treating physician

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-10; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects achieving a 13mm or more reduction in pain as measured on a 100-mm VAS within 30 minutes. | 30 minutes

SECONDARY OUTCOMES:
Median maximum reduction in VAS pain score achieved within 30 minutes | 30 minutes
Median time required to achieve a 13-mm reduction in VAS pain score | 1 hour
Vital signs changes (ETCO2, O2sat, HR, RR, BP) | 1 hour
  Changes in vital signs will be recorded every 5 minutes for 30 minutes, then every 10 minutes for 30 minutes
Adverse effects as defined by SERSDA | 1 hour
  SERSDA (Side Effect Rating Scale for Dissociative Anaesthesia) includes: fatigue, dizziness, nausea, headache, feeling of unreality, changes in hearing, changes in vision, mood change, generalized discomfort, and hallucination.

CONTACTS AND LOCATIONS:
Overall Officials: Gary Andolfatto, MD, Principal Investigator — UBC Dept of EM; Lions Gate Hospital
Locations (1):
- Lions Gate Hospital, North Vancouver, British Columbia, Canada